CLINICAL TRIAL: NCT04293263
Title: The Effect of Shared Listening to Personalized Music on Symptoms of Behavioral Disorders in the Elderly With Advanced Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: 2gether (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2020-02-16; First posted 2020-03-03 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Dementia
Keywords: music therapy
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCI patients hospitalised in the research departments (Experimental): each of the elderly in the study group will listen to personalized music twice a week for an hour each time together with a musical partner. Joint listening is performed with 2 pairs of headphones that connect via a splitter to the partner's cell phone. A listening session will take place in a period of 30 minutes and not more than 60 minutes.
  Interventions: Combination Product: 2gether app used by trained personal
- MCI patients hospitalized in the research departments (Active Comparator): each of the elderly in the control group will Listen to random music twice a week for about 40 minutes each time, on personal headphones.
  Interventions: Combination Product: 2gether app used by trained personal

INTERVENTIONS:
Combination Product: 2gether app used by trained personal — each of the elderly in the study group will listen to personalized music twice a week for an hour each time together with a musical partner. Joint listening is performed with 2 pairs of headphones that connect via a splitter to the partner's cell phone. A listening session will take place in a period of 30 minutes and not more than 60 minutes.
  Musical partner - A person trained in the program's work plan, which includes contact with empathic listening and the use of a dedicated application developed for it. A musical partner will meet with the same elderly person throughout the study period.
  Empathetic listening - a situation in which a person listens to music with another person, while the music enables contact and deepening the connection between people.
  Other Names: Listen to random music twice a week for about 40 minutes each time, on personal headphones.

SUMMARY:
This study is of great importance because it uses a method that has not been tested in the past. To date, various interventions have been examined that use music for patients with dementia. At the same time, no intervention was conducted that integrates an additional person who shares personalized music with the patient.

If the combination of another person who shares the positive effect of the music with the patient is found to enhance the positive effect of the music, it can change the routine of work with dementia patients and may even reduce the use of tranquilizers among them.

In many cases, it has been found that one of the biggest challenges for family members who treat patients with dementia is the lack of content in the sessions and as a result, the growing sense of alienation between the patient and his family.

Listening to music can be a significant tool in the hands of the family, the main caregiver, the medical staff, and any person who comes in contact with the patient, a tool that can strengthen the sense of connection and connection between them.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the Department of Mental Disorders at the Mental Health Center in Be'er Sheva aged 18 and over.
* Patients who have been diagnosed with dementia for the issue.
* Patients whose guardian gave consent for the study.

Exclusion Criteria:

* Hearing-impaired patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
change in BPSD measure among patients in the department. we use the Neuropsychiatric Inventory (NPI) (Cummings et al., 1994.) which detects changes in BPSD. | 8 month
  the measured scale estimates 10 out of 12 common behavioural disorders in Dementia: delusions, hallucinations, depression, anxiety, agitation, aggression, euphoria, inhibitions, irritability or instability, , Abnormal motor activity. A higher score indicates a larger severity of these behaviours. min-0 max-140. The follow-up will be performed by a nurse in both departments on a weekly basis during 8 months of the study.

SECONDARY OUTCOMES:
change in the professional caregivers impression of the treatment | 8 month
  We will use a global improvement subclass. This is a scale of 7 points, "1" - the situation has improved greatly and "7" - the situation has worsened greatly.
change vigor measures of the department's staff (nursing staff) | 8 month
  burnout is a common challenge among caregivers of dementia patients. we use Shirom-Melamed Vigor Measure (SMVM) tool. a 12-item tool with a minimum score indicating a higher incidence of wear.

IPD SHARING:
Plan to Share IPD: Undecided